CLINICAL TRIAL: NCT01402297
Title: Hydrogen Peroxide and Nitrite Reduction in Exhaled Breath Condensate of COPD Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Collaborators: Ministry of Science and Higher Education, Poland (Other Government)
Responsible Party: Medical University of Lodz, Medical University of Lodz, Lodz, Poland
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Nowak-02
Record Dates: First submitted 2011-07-18; First posted 2011-07-26 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: apocynin; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — acetovanillone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- COPD patients (Experimental): Thirteen nonsmoking patients, suffering from GOLD II and GOLD III stage participated in the study (mean age 57 years (range 42-79), 9 men, 4 women). COPD was diagnosed based on GOLD 2009 criteria. All the participants were diagnosed at Department of Clinical Physiology, Medical university of Lodz.
  Interventions: Drug: Apocynin and placebo nebulization

INTERVENTIONS:
Drug: Apocynin and placebo nebulization — 6 ml of apocynin of total dose 3 mg (0.5 mg/ml dissolved in sterile 0.9% NaCl as the study drug) and 0,9% NaCl as placebo, has been nebulized for 15-20 min through the mouthpiece with using of a nose clip. A nebulizer Pulmo Aide AP-50 (DeVilbiss; Richmond, VA) was used (mass median aerosol diameter 3.1 mm, output 0.3 ml/min.)
  Other Names: 4-hydroxy-3-methoxyacetophenone,; acetovanillone

SUMMARY:
The aim of the study is to investigate the effect of inhaled apocynin on ROS (reactive oxygen species) and NOS (reactive nitrogen species) synthesis in 13 COPD patients. Effects of nebulized apocynin (0.5 mg/ml, 6 ml) were assessed in exhaled breath condensate (EBC) after 30, 60 and 120 minutes.

DETAILED DESCRIPTION:
Apocynin reduced hydrogen peroxide concentration in exhaled breath condensate 60 and 120 minutes after apocynin nebulization comparing to placebo (0.43 μM vs. 0.59 μM and 0.41 μM vs. 0.58 μM respectively, p<0.05). Interestingly, apocynin caused decrease of NO2- concentration 30, 60 and 120 minutes after apocynin inhalation (3.9 μM vs. 4.5 μM, 3.8 μM vs. 4.5 μM and 3.7 μM vs. 4,4 μM respectively, p<0.05) comparing to placebo, but did not cause any significant changes in concentration of NO3- in any timepoint (p>0.05). No influence of apocynin on safety parameters, and no adverse effects has been observed.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from bronchial COPD (II and III stage)
* patients free of any medication few days before research
* patients had not suffered from any infectious diseases including upper respiratory tract infections for at least 3 months prior to the study

Exclusion Criteria:

* Patients suffering from GOLD I stage
* patients taking medications few days before the study
* infectious diseases that had occurred 3 months or less before the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 3 months
  Apocynin Did Not Cause Any Adverse Effect or influence blood pressure
Peripheral Blood Differential Count | 3 months
  Apocynin did not influence Peripheral Blood Differential Count and did not cause any adverse events
Lung function tests (spirometry) | 3 months
  Apocynin did not cause changes in lung function tests
Single Breath Carbon Monoxide Diffusing Capacity (DLCO) | 3 months
  Single breath DLCO was not modified by apocynin nebulization.

SECONDARY OUTCOMES:
Determination of H2O2 | 3 months
  apocynin decreased H2O2 concentrations 60 and 120 minuter after nebulization in comparison to placebo
Determination of NO3- concentration in Exhaled Breath Condensate | 3 months
  Apocynin did not influence NO3- concentration in Exhaled Breath Condensate
Determination of NO2- concentration in Exhaled Breath Condensate | 3 months
  Apocynin decreased NO2- concentration in Exhaled Breath Condensate 30, 60 and 120 minuter after nebulization in comparison to placebo
Determination of NO2- Concentration in Serum | 3 months
  No influence of apocynin on NO2- Concentration in Serum was observes
Blood Pressure | 3 months
  No influence of apocynin on blood pressure was observed
Peripheral Blood Differential Count | 3 months
  Apocynin Did Not Cause Any Adverse Effect or influence Peripheral Blood Differential Count
Lung Functional Tests | 3 months
  Single breath DLCO was not modified by apocynin nebulization.
Single Breath Carbon Monoxide Diffusing Capacity (DLCO) | 3 months
  Apocynin did not influence DLCO

CONTACTS AND LOCATIONS:
Overall Officials: Rafal Pawliczak, Professor, Study Chair — Medical University of Lodz